CLINICAL TRIAL: NCT04225793
Title: Comparative Analysis of the Osmotic Laxative Application Efficiency and Safety Eziclen and Moviprep for Colonoscopy Preparation
Brief Title: The Use of Osmotic Laxatives Versus Macrogol for Bowel Preparation in Patients Undergoing Colonoscopy
Acronym: CLEAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 685476
Record Dates: First submitted 2019-10-24; First posted 2020-01-13 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Disorders
Keywords: colorectal cancer; colonoscopy; Eziclen
MeSH Terms: conditions — Colorectal Neoplasms | interventions — formyldienolone; MoviPrep; Polyethylene Glycols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eziklen® (Active Comparator): potassium, magnesium and sodium sulphates-based laxative
  Interventions: Drug: Eziklen®
- Macrogol (Active Comparator): Macrogol-3350 + Sodium Sulfate + Potassium Chloride+ Sodium Chloride + Ascorbic Acid-based and Sodium Ascorbate-based Moviprep
  Interventions: Drug: MoviPrep

INTERVENTIONS:
Drug: Eziklen® — The Eziclen solution should be taken in the one-time use regimen in morning before procedure.
  Consumption of the full volume of the Eziklen® solution of the preparation and the additional amount of water or a clear liquid should be completed at least 2 hours and no later than 4 hours before the procedure.
  Other Names: esiclene, Eziklen
  Arms: Eziklen®
Drug: MoviPrep — The Moviprep® solution should be taken in the one-time use regimen in morning before procedure.
  Consumption of the full volume of the Moviprep® solution should be completed at least 2 hours and no later than 4 hours before the procedure.
  Other Names: Moviprep, macrogol
  Arms: Macrogol

SUMMARY:
The gold standard of colorectal examination is colonoscopy. One of the main purposes of colonoscopy is detecting bowel neoplasms. Right now there are several methods the bowel preparation for the colonoscopy.

Several factors can affect the quality of the bowel preparation, such as the kind of oral laxative, the time after its intake and the diet followed in the days before colonoscopy. In this randomized clinical trial the investigators aimed to compare the safety and efficiency of two low-volume laxatives for bowel preparation: potassium, magnesium and sodium sulphates-based laxative Eziclen (IPSEN, France) and Macrogol-3350 + Sodium Sulfate + Potassium Chloride+ Sodium Chloride + Ascorbic Acid-based and Sodium Ascorbate-based Moviprep (Nordgine B.V., The Netherlands)

DETAILED DESCRIPTION:
The key method of colorectal examination is colonoscopy. The result, diagnostic significance and therapeutic safety depend a lot on the quality of bowel preparation. One of the main purposes of colonoscopy is detecting the earliest forms of colorectal cancer and prognostically meaningful small nonpolyposis neoplasms. The good and perfect bowel preparation is essential in this case.

However, the bowel preparation for colonoscopy must fulfill the following criterias:

* Be effective, that means to empty colon of faeces, residual liquid and foamy content fully and safely;
* Harmless, no side effects on the other organs and systems;
* Do not cause discomfort nor change to electrolyte balance, well tolerated;
* Do not affect the severity of bowel disease nor cause macro- and microscopic colon mucose changes;
* Quick response with short preparation period (no more than 24 hours);
* Easy to use, so patient could perform it independently or with the least medical staff participation;
* Do not require special conditions, equipment and staff training (possibility to perform at home);
* Do not distort the endoscopic image (colour, shape, reflexion);
* Do not limit the use of vital dyes or other means of endoscopic diagnosis and treatment;
* Do not damage the endoscopic equipment;
* be cheap . Bowel preparation schemes usually include diet (low-residue) and oral laxative intake. The low-residue diet should last no more than 24 hours before the colonoscopy according to the European Society of Gastrointestinal Endoscopy clinical recommendations.

The time factor is essential for quality of bowel preparation. If the colonoscopy is performed in the first half of day the intake of the part of laxatives (usually a half) on that day (split-mode or separate) provides a better result in comparison to full dose intake on the colonoscopy day or the evening before it.

Bowel preparation might be fully undertaken (in full volume) in the morning of examination day for patients undergoing colonoscopy in the afternoon according to some studies. In the case of laxative intake on the morning of examination day, excellent preparation quality and good patient tolerance was demonstrated in the Varughese S et al. research assessing 4 liters bowel preparation scheme efficiency for patients undergoing colonoscopy in the afternoon in comparison to intake in the evening before colonoscopy.

The patient's somatic status and the urgency should be considered for choosing the bowel preparation mode.

Polyethyleneglycol-based drugs have become more commonly used in clinical practice for colonoscopy bowel preparation since its appearance in 1980.

The drug passes through the intestine without being absorbed and metabolized and increases the bowel liquid volume, as do all osmotic laxatives. Thus, electrolyte balance is not disrupted and effective intestinal lavage occurs. But patient compliance might be influenced significantly due to a large volume intake requirement (4 l) and specific organoleptic feature.

Over the course of several years, European and Canadian experts have accepted the sodium picosulfate+ magnesium citrate-based low-volume bowel preparation method (2l) as alternative option and the FDA has also approved it in July 2012.

This combined intake scheme allows to prepare intestine efficiently for the examination. The sodium picosulfate has a bowel stimulating effect and as osmotic laxative magnesium citrate retains water. But the electrolyte balance changes and dehydration may also influence the patient compliance to laxative.

According to the international clinical recommendations for colonoscopy, 4l polyethylenуglycol-based laxative in split-mode preparation with an time interval no more than 4 hours from the end of preparation until colonoscopy is recommended as a standard method. Low-dose polyethylenуglycol-based laxative intake (2l) combined with ascorbate or sodium thiosulfate+ magnesium citrate can serve as alternative examination preparation method (especially for outpatients). Only polyethylenуglycol-based laxative can be recommended for patients with renal failure as bowel preparation method.

Eziclen - potassium, magnesium and sodium sulphates-based osmotic laxative for colonoscopy preparation registered in Russia doesn't have a strong evidence base and is not included in national recommendations yet due to its recent market entry (2018) But according to the registered multicenter controlled clinical trials assessing the potassium, magnesium and sodium sulfates vs. 2l polyethyleneglycol with electrolytes efficiency for colonoscopy preparation in split-mode (n=356) and one-day preparation (n=364) (primary endpoint - bowel purity degree as "perfect", "good", "bad") as well as non-conceded Eziclen efficiency was identified in comparing to the control group (97,2% vs 96,1% and 84% vs 82,9% respectively). The side effects frequency was also comparable with control group. There was shown a comparable rate of effective bowel preparation (97,2% vs 97,7%) on a background of higher patient compliance (95,7 % comparing to 82,3 %) in a similar study assessing Eziclen efficiency, safety and patient compliancy in comparison with Macrogol 400 with electrolytes.

So the investigators aimed our study to investigate efficiency, safety and compliance of two low-volume laxatives Potassium Sulfate+ Magnesium Sulfate+ Sodium Sulfate-based (Eziclen) vs. relevant volume of Macrogol-3350+ Sodium Sulfate+ Potassium Chloride+ Sodium Chloride+ Ascorbic Acid and Sodium Ascorbate-based (Moviprep) in bowel preparation for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent forms confirming the understanding of the course of study and agreement to participate in it.
2. A written patient consent to fill the prepared questionnaire and to perform diagnostic colonoscopy in case of following situations:

   * Routine oncological screening
   * Polyps or neoplasms in anamnesis
   * Anemia or latent bleeding diagnostics
   * Diarrhea or constipation with unknown reason
   * Inflammatory bowel disease in remission
   * Pathological formation according to US examination (neoplasm evidence in abdomen)
3. Suspicious colon neoplasms according to CT and/or irrigography
4. ASA scale for physical status assessment ≤ 3
5. Patients with adequate electrolyte balance rate (K, Na, Cl, bicarbonate rate screening).

Non-inclusion criteria:

1. The baseline data about comorbidities or laboratory data that can jeopardize the safety of the patient or reduce the likelihood of obtaining satisfactory data necessary to achieve the goal (goals) of the study.
2. The presence of progressive carcinoma or other bowel disease, leading to excessive mucous membrane fragility.
3. The confirmed or suspected gastrointestinal (FA) obstruction, stagnation in the stomach, gastroparesis, or a violation of gastric evacuation.
4. The intestinal perforation.
5. The profuse vomiting.
6. The procedure goal to perform a medical procedure (eg, polypectomy, mucosectomy).
7. The presence of toxic colitis or megacolon.
8. Severe acute phase of inflammatory bowel disease as a contraindication to colonoscopy.
9. The presence of acute GI bleeding.
10. History of gastrointestinal surgery (for example, colostomy, colectomy, gastric bypass surgery, stomach resection).
11. The history of impaired consciousness predisposing to pulmonary aspiration.
12. The colonoscopy aimed remove a foreign body or decompression.
13. History of incomplete colonoscopy
14. The confirmed severe renal failure (glomerular filtration rate (GFR) <30 ml / min / 1.73 m2).
15. The confirmed severe liver failure (10-15 points on the Child-Pugh scale).
16. Dehydration condition requiring treatment.
17. The ascites.
18. Severe congestive heart failure (class III and IV).
19. The state of hyperuricemia with a clinic of gouty arthritis.
20. Pregnancy or lactation.
21. Patients at risk of pregnancy and not using an acceptable method of contraception during the study. Women of childbearing age must provide a negative pregnancy test at the beginning of the study and must use the oral contraceptive method, double (use a condom with spermicidal gel, birth control suppositories or films; diaphragm with spermicides; or male condom and diaphragm with spermicides), injection contraception or intrauterine devices . Non-fertile women - more than a year after menopause, after surgical sterilization or hysterectomy at least 3 months before the start of the study.
22. The hypersensitivity reaction to active substances or to other auxiliary substances (Eziklen and Moviprep).
23. A patient with a mental state that does not allow him to understand the nature, extent and possible consequences of the study and / or evidence of refusal to cooperate.
24. During the course of the study, the patient is likely to require treatment with drugs that are not permitted by the study protocol.

Exclusion Criteria:

1. The pregnancy
2. The inability to follow the protocol
3. Refuse of study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2020-06-02 (Estimated); Study Completion 2020-08-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of bowel preparation according to Boston Bowel Preparation Scale | during the procedure
  Total score of bowel preparation measured from 0 to 9. The maximum BBPS score for a perfectly clean colon without any residual liquid is 9 and the minimum BBPS score for an unprepared colon is 0. This is evaluated by the endoscopist

SECONDARY OUTCOMES:
Patient compliance to preparation | 1 houre before procedure
  is measured with a specially designed questionnaire, 4 points, where 0 is very use it again and 4 will advise to all
adverse events rate | starting 1 day before the procedure and within 2 weeks after
  is measured as from 0 to 4 in case of presence any complication (nausea or vomiting or headache or abdominal pain related to preparation)
The polyps detection rate | during the procedure
  is measured as 0 in cases there were no polyps or 1 in case if there were polyps detected by colonoscopy
Researcher satisfaction with preparation | during the procedure
  Satisfaction of the operator will be evaluated on a 5-point Likert scale with a range from 0 to 4 points, where 0 is insufficient and 4 complete bowel preparation.
sodium blood level | one the day before procedure and one houre before procedure
  mg per ml
potassium blood level | one the day before procedure and one houre before procedure
  tmg per ml
creatinine blood level | one the day before procedure and one houre before procedure
  mg per dl
urea blood serum level | one the day before procedure and one houre before procedure
  mg per ml

CONTACTS AND LOCATIONS:
Overall Officials: Inna Tulina, PhD, Study Director — Russian Society of Colorectal Surgeons; Pavel Pavlov, PhD, Study Chair — Russian Society of Colorectal Surgeons; Andrey Kiryukhin, Principal Investigator — Sechenov State University
Locations (1):
- Clinic of Colorectal and Minimally invasive surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No